CLINICAL TRIAL: NCT02893241
Title: Cafedrin/Theodrenalin (Akrinor®) Versus Ephedrine for Treatment of Hypotension in the Peri-operative Phase in Inpatient Setting: a Multicenter, Prospective, Non-interventional Study
Brief Title: Cafedrin/Theodrenalin (Akrinor®) Versus Ephedrine for Treatment of Hypotension in the Peri-operative Phase in Inpatient Setting
Status: Completed | Type: Observational
Sponsor: Ratiopharm GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: TV48531-CV-40092
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — cafedrine, theodrenaline drug combination; Ephedrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Patients ≥ 50 years old, with pre-existing comorbidities, who receive general anaesthesia
  Interventions: Drug: Cafedrine/theodrenaline; Drug: Ephedrine
- Cohort B: Patients, who undergo caesarean section under spinal anaesthesia
  Interventions: Drug: Cafedrine/theodrenaline; Drug: Ephedrine

INTERVENTIONS:
Drug: Cafedrine/theodrenaline
Drug: Ephedrine

SUMMARY:
This is a national, multicentre, prospective, open, two-arm, non-interventional study with hospitalized patients, who are treated routinely with cafedrine/theodrenaline or ephedrine after occurrence of perioperative hypotension, wherein the patients are assigned to a treatment arm based on the department.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients, who received IV treatment (bolus administration) with cafedrine/theodrenaline or ephedrine (Ephedrin Meduna) due to an acute arterial hypotension
* Consent to use of data is available
* Patient under careful blood pressure and pulse monitoring (at least 2 minutes measuring interval (BP/HR) and/or at least 7 measurements within the first 15 minutes after the first application of cafedrine/theodrenaline or ephedrine)

Cohort A:

* Treatment of hypotension in < 100 mm Hg syst. and/or drop in blood pressure > 20% syst. compared to preoperative base value (syst.)
* Patients ≥ 50 years old
* Pre-existing comorbidities (ASA classification 2-4)
* Elective surgery
* General anaesthesia with propofol/fentanyl ≥ 0.2 mg (or equivalent)

Cohort B:

* Treatment of hypotension in < 100 mm Hg syst. and/or drop in blood pressure > 10% syst. compared to preoperative base value (syst.)
* Patients ≥ 18 years old
* Caesarean section under spinal anaesthesia

Exclusion Criteria:

* Contraindication to the use of cafedrine/theodrenaline or ephedrine (Ephedrin Meduna) in accordance with current German specialist information

  * Hypersensitivity to any product ingredient
  * Hypertensive blood pressure readings
  * Mitral stenosis
  * Narrow-angle glaucoma
  * Hyperthyroidism
  * Pheochromocytoma
  * Prostatic adenoma with urinary retention
  * Bronchial asthmatics with sulphite sensitivity
  * Hyper-excitability
  * Arteriosclerosis
  * Aneurysm
  * Treatment with other indirect sympathomimetic drugs (Example: phenylpropanolamine, phenylephrine, pseudoephedrine or methylphenidate)
  * Use of Monoamine oxidase (MAO) inhibitors (including within the last two weeks)
* Prophylactic administration of cafedrine/theodrenaline or ephedrine or other anti-hypertensives
* Sepsis, septic shock or systemic inflammatory response syndrome (SIRS)

Cohort A:

• Intra-cranial surgery or heart surgery

Cohort B:

* High-risk pregnancy (emergency Caesarean, severe infantile malformation)
* Multiple pregnancy
* Amniotic infection syndrome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hospitalized patients, who are treated routinely with cafedrine/theodrenaline or ephedrine after occurrence of perioperative hypotension,
Sampling Method: Non-Probability Sample
Enrollment: 2013 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of newly occurring HR ≥ 100 beats/min | during the first 15 minutes after initial drug administration of cafedrine/theodrenaline or ephedrine
Weighted deviation below the individually determined, lowest systolic blood pressure BPmin | within the first 15 minutes after the initial delivery of the antihypotonic drug as area1 (AUC) between the systolic blood pressure curve (below BPmin) and the lower limit BPmin

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (75):
- Germany (75):
  - Teva Investigational Site 133, Aachen
  - Teva Investigational Site 122, Amberg
  - Teva Investigational Site 106, Aue
  - Teva Investigational Site 116, Augsburg
  - Teva Investigational Site 165, Aurich
  - Teva Investigational Site 110, Bad Hersfeld
  - Teva Investigational Site 134, Bad Saarow
  - Teva Investigational Site 174, Bad Soden
  - Teva Investigational Site 142, Baden-Baden
  - Teva Investigational Site 121, Brake
  - Teva Investigational Site 146, Cologne
  - Teva Investigational Site 154, Dillingen
  - Teva Investigational Site 119, Dresden
  - Teva Investigational Site 171, Düsseldorf
  - Teva Investigational Site 111, Eichstätt
  - Teva Investigational Site 107, Essen
  - Teva Investigational Site 167, Flensburg
  - Teva Investigational Site 141, Friedberg
  - Teva Investigational Site 131, Fulda
  - Teva Investigational Site 114, Gelnhausen
  - Teva Investigational Site 158, Gelsenkirchen
  - Teva Investigational Site 164, Giessen
  - Teva Investigational Site 149, Göppingen
  - Teva Investigational Site 159, Greifswald
  - Teva Investigational Site 113, Hamburg
  - Teva Investigational Site 163, Hamburg
  - Teva Investigational Site 143, Hanover
  - Teva Investigational Site 144, Hanover
  - Teva Investigational Site 151, Hanover
  - Teva Investigational Site 129, Heilbronn
  - Teva Investigational Site 112, Herford
  - Teva Investigational Site 160, Hildesheim
  - Teva Investigational Site 132, Homburg
  - Teva Investigational Site 168, Idar-Oberstein
  - Teva Investigational Site 147, Jena
  - Teva Investigational Site 123, Karlsruhe
  - Teva Investigational Site 157, Kassel
  - Teva Investigational Site 104, Kempen
  - Teva Investigational Site 117, Leipzig
  - Teva Investigational Site 135, Leipzig
  - Teva Investigational Site 118, Leverkusen
  - Teva Investigational Site 102, Lingen
  - Teva Investigational Site 109, Ludwigsburg
  - Teva Investigational Site 139, Lüneburg
  - Teva Investigational Site 101, Marburg
  - Teva Investigational Site 155, Minden
  - Teva Investigational Site 138, Mönchengladbach
  - Teva Investigational Site 127, München
  - Teva Investigational Site 130, Münster
  - Teva Investigational Site 124, Neuruppin
  - Teva Investigational Site 152, Nuremberg
  - Teva Investigational Site 173, Nuremberg
  - Teva Investigational Site 156, Oldenburg
  - Teva Investigational Site 108, Pforzheim
  - Teva Investigational Site 136, Pirmasens
  - Teva Investigational Site 172, Prien am Chiemsee
  - Teva Investigational Site 150, Rheine
  - Teva Investigational Site 125, Rostock
  - Teva Investigational Site 169, Saalfeld
  - Teva Investigational Site 148, Schwalmstadt
  - Teva Investigational Site 166, Schwerin
  - Teva Investigational Site 126, Solingen
  - Teva Investigational Site 128, Traunstein
  - Teva Investigational Site 170, Trier
  - Teva Investigational Site 175, Ulm
  - Teva Investigational Site 162, Unna
  - Teva Investigational Site 153, Velbert
  - Teva Investigational Site 105, Warendorf
  - Teva Investigational Site 115, Wesel
  - Teva Investigational Site 140, Wetzlar
  - Teva Investigational Site 120, Wiesbaden
  - Teva Investigational Site 137, Worms
  - Teva Investigational Site 103, Würzburg
  - Teva Investigational Site 145, Zwiesel
  - Teva Investigational Site 146, Zwiesel

REFERENCES:
- [Derived] Kranke P, Geldner G, Kienbaum P, Gerbershagen HJ, Chappell D, Wallenborn J, Huljic S, Koch T, Keller T, Weber S, Kunitz O, Linstedt U, Eberhart LHJ; HYPOTENS study group. Treatment of spinal anaesthesia-induced hypotension with cafedrine/theodrenaline versus ephedrine during caesarean section: Results from HYPOTENS, a national, multicentre, prospective, noninterventional study. Eur J Anaesthesiol. 2021 Oct 1;38(10):1067-1076. doi: 10.1097/EJA.0000000000001474. PMID 33625060
- [Derived] Eberhart L, Geldner G, Huljic S, Marggraf K, Keller T, Koch T, Kranke P. A non-interventional comparative study of the 20:1 combination of cafedrine/theodrenaline versus ephedrine for the treatment of intra-operative arterial hypotension: the 'HYPOTENS' study design and rationale. Curr Med Res Opin. 2018 Jun;34(6):953-961. doi: 10.1080/03007995.2018.1438379. Epub 2018 Feb 28. PMID 29415580